CLINICAL TRIAL: NCT06313034
Title: The Effect of Breastfeeding Training for Mothers Who Have a Vaginal Birth With Motivational Interview Technique on Their Breastfeeding Motivation, Self-efficacy, and Attachment
Brief Title: The Effect of Breastfeeding Training Given to Mothers With Vaginal Birth by Motivational Interview Technique
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gümüşhane Universıty (Other)
Collaborators: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Özge PALANCI AY, Principal Investigator, Gümüşhane Universıty
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GU-SBF-OPA-02
Record Dates: First submitted 2024-03-05; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Breastfeeding
Keywords: Attachment; Breastfeeding Motivation; Breastfeeding Self-Efficacy; Mother; Motivational Interview
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: The sample of the research will consist of mothers who gave primary vaginal birth (40 experimental group and 40 control group)
Who Masked: Participant
Masking Description: While it is known by the researcher whether the mothers are in the experimental or control group, it is not known by the mother.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Breastfeeding education will be given to mothers in the experimental group in 4 individual and face-to-face sessions based on motivational interviewing technique.
  The first session of breastfeeding training based on motivational interviewing technique will be held in the delivery room where the mother is hospitalized before being discharged from the hospital. Other sessions will be held according to the monitoring frequency recommended in the Postnatal Care Management Guide of the Ministry of Health of the Republic of Turkey (2018). These will be done at the health institution where the mother receives service.
  Second session; Between the 2th and 5th postpartum day Third session; Between the 13th and 17th postpartum day Fourth session; Between the 30th and 42th postpartum day The duration of each motivational interview is planned to be between 30-40 minutes on average.
  Interventions: Behavioral: Breastfeeding education based on motivational interviewing technique
- control group (No Intervention): Before discharge, mothers in the control group will be given routine breastfeeding training by the midwife working in the delivery room in accordance with the mother/baby friendly hospital protocol.

INTERVENTIONS:
Behavioral: Breastfeeding education based on motivational interviewing technique — Breastfeeding education based on motivational interviewing technique; Breast milk properties, benefits to mother and baby, breastfeeding positions, the relationship between breastfeeding and attachment, signs of hunger in the newborn, Breastfeeding frequency, duration and termination, Breast milk expressing methods, Expressions showing that the newborn has enough milk, Breast milk storage will cover the topics. These topics will be given based on motivational interviewing technique.
  According to the motivational interviewing technique, the mother's "intention, importance and confidence-sufficiency" regarding breastfeeding will be determined and firstly, an agenda will be created on "issues related to breastfeeding with the mother". Each session will be conducted by following the "open-ended questioning, verification, reflective listening and summarizing" approaches of the motivational interviewing technique.
  Arms: experimental group

SUMMARY:
This study aimed to determine the effect of breastfeeding education given to mothers who gave birth vaginally using motivational interviewing technique on breastfeeding motivation, self-efficacy and attachment. The study will be conducted as a single-blind, randomized controlled trial.

DETAILED DESCRIPTION:
The study will be conducted as a single-blind, randomized controlled trial with 80 mothers who gave birth vaginally. In the experimental group, just before discharge from the hospital (within the last 4 hours before discharge), on the 2nd-5th, 13th-17th, 30th-42nd days after birth. Breastfeeding training based on motivational interviewing technique will be given 4 times in total. The control group will continue to receive the current standard care and service of the relevant hospital and other postpartum health institutions.

Hypotheses of the Research

1. The effect of breastfeeding education given to mothers who gave birth vaginally with motivational interviewing technique on increasing the mother's breastfeeding motivation.

   are there?(H1)
2. Breastfeeding education given to mothers who gave birth vaginally with motivational interviewing technique has no effect on increasing the mother's breastfeeding self-efficacy.

   Does it have any effect?(H2)
3. The effect of breastfeeding education given to mothers who gave birth vaginally with motivational interviewing technique on increasing the level of mother-infant attachment.

are there?(H3)

ELIGIBILITY:
Inclusion Criteria:

Maternal criteria;

* Agreeing to participate in the research
* Being 20 years or older
* Having had a vaginal birth
* being primiparous
* Being at least a primary school graduate
* Ability to speak Turkish
* Not having any condition that would prevent communication
* No medical breast problem

Criteria for the baby;

* Being born at term (38-41 gestational weeks)
* There is no congenital anomaly such as cleft palate or lip of the newborn that may prevent sucking.
* Birth weight over 2500 grams

Exclusion Criteria:

Maternal criteria;

* Having a chronic disease that prevents breastfeeding
* Having major breast problems that will prevent breastfeeding
* The mother has a diagnosed psychiatric disease
* Having 2 or more live newborns in this birth

Criteria for the baby;

* Premature birth (37th gestational week and before)
* Having a congenital disease
* Being in the risk group/being diagnosed with a disease in the newborn screening program

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-03-15 (Estimated); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
Mother Introductory Information Form | one day
  It was prepared in line with the literature. The form consists of a total of 27 questions, including information about socio-demographic information, obstetric, newborn characteristics.breastfeeding characteristics
Primipara Breastfeeding Motivation Scale | Three months
  It was developed to determine the factors affecting breastfeeding motivation in primiparous women. The scale is a 7-point Likert type, consisting of a total of 29 items and 4 sub-dimensions. These sub-dimensions; the value placed on breastfeeding, self-efficacy, perceived midwife support and expectation of success. There is no cut-off value and total score in the evaluation of the scale. As the score obtained from each sub-dimension increases, the breastfeeding motivation level of that sub-dimension increases.
Breastfeeding Self-Efficacy Scale Short Form | Three months
  The scale is a 5-point Likert type and consists of 14 questions in total. The lowest score that can be obtained from the scale is 14 and the highest score is 70. High scores are interpreted as high breastfeeding self-efficacy.
Mother-Baby Attachment Scale | Three months
  The scale has a total of 8 items and is a 4-point Likert type. Responses are scored between 0-3. In the evaluation, items with positive emotion expressions (1, 4, 6.) were scored as 0, 1, 2, 3, while items with negative emotion expressions (2, 3, 5, 7, 8.) were scored as 3, 2, 1,0. It is scored as. The lowest score that can be obtained from the scale is 0 and the highest score is 24. As the score obtained from the scale increases, the level of mother-infant attachment decreases

CONTACTS AND LOCATIONS:
Overall Officials: ÖZGE PALANCI AY, Principal Investigator — Gümüşhane Universıty; SONGÜL AKTAŞ, Principal Investigator — Karadeniz Technical University
Locations (1):
- Gümüşhane University, Gümüşhane, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No